CLINICAL TRIAL: NCT02647827
Title: Acupuncture or Metformin for Insulin Resistance in Women With Polycystic Ovary Syndrome: A Randomized Controlled Trial
Brief Title: Acupuncture or Metformin for Insulin Resistance in Women With PCOS
Acronym: PIAII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Peking University (Other)
Responsible Party: Principal Investigator, Elisabet Stener-Victorin, PhD, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT: 2015-004250-18; 2015-004250-18 (EudraCT Number)
Record Dates: First submitted 2015-12-23; First posted 2016-01-06 (Estimated); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Polycystic Ovary Syndrome; Insulin Resistance; Hyperandrogenism
Keywords: Acupuncture; Metformin; Glucose metabolism; Hba1c
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Hyperandrogenism | interventions — Acupuncture Therapy; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lifestyle management (Active Comparator): All women will receive lifestyle management instructions at the baseline visit, before randomization.
  Interventions: Other: Lifestyle management
- Acupuncture + lifestyle management (Active Comparator): Three treatment per week (4 weeks) and thereafter 2 times per week during 12 weeks.
  Interventions: Other: Lifestyle management; Device: Acupuncture
- Metformin + lifestyle management (Active Comparator): Oral metformin 500 mg three times daily, in total 1500 mg per day.
  Interventions: Other: Lifestyle management; Drug: Metformin

INTERVENTIONS:
Other: Lifestyle management — All women will receive lifestyle management instructions at the baseline visit, before randomization. The lifestyle management involves one initial counselling session in connection with the baseline visit, which includes information about the importance of weight management, healthy diet and physical activity.
Device: Acupuncture — Disposable, single-use, sterilized CE marked needles made of stainless steel, 0.25 x 30 mm and 0.30 x 40/50 mm will be inserted to a depth of 15-40 mm in segmental acupuncture points located in abdominal and leg muscles, with innervations corresponding to the ovaries and the pancreas. Two sets of acupuncture points will be alternated every second treatment.
  Arms: Acupuncture + lifestyle management
Drug: Metformin — Oral metformin 500 mg three times daily, in total 1500 mg per day. To reduce gastrointestinal side-effects of metformin, the dose will be slowly escalated starting with 500 mg daily during the first week, increasing to 500 mg twice per day during the second the week, and 500 mg three times daily, morning, lunch and dinner from the third week in total 16 weeks including the 3 weeks step-up phase (i.e. 4 months).
  Arms: Metformin + lifestyle management

SUMMARY:
The hypothesis is that acupuncture is equally effective as metformin (both treatments combined with lifestyle management) in improving whole body glucose homeostasis in insulin resistant women with polycystic ovary syndrome (PCOS), and that both are superior to lifestyle management alone. The investigators hypothesize that acupuncture and metformin induce ovulation and improve hyperandrogenism, as well as health related quality of life (HRQoL) and symptoms of anxiety and depression. Although equally effective (acupuncture and metformin), the investigators hypothesize that acupuncture is associated with less negative side-effects. The investigators also hypothesize that these treatments have the potential to restore epigenetic and molecular alterations in target tissues (endometrial-, adipose-, and skeletal muscle tissue) and thus have the potential to prevent the development of type 2 diabetes (T2D).

DETAILED DESCRIPTION:
Specific Aims The purpose of the study is to perform a randomized controlled trial of women with PCOS, comparing the effectiveness of lifestyle management alone, and in combination with acupuncture or metformin treatment on whole body glucose homeostasis, with the ultimate goal to prevent the development of type 2 diabetes.

Primary aim

1. To determine the clinical effectiveness of 4 months of 1) electroacupuncture + lifestyle management and 2) metformin + lifestyle management, compared to 3) lifestyle management only, for improvement of insulin sensitivity as measured by HOMA-IR, by the insulin response to glucose assessed by calculating the area under the curve (AUCinsulin) during the oral glucose tolerance test (OGTT), and by glucose regulation (assessed by analyzing Hba1c levels).

Secondary aims

1. To evaluate changes in secondary metabolic measures, including fasting insulin, c-peptide, glucose, and adipokines, calculation of HOMA-B (i.e. the Islet β-cell function) and the c-peptide index, assessment of the adipokines and lipid profile, body size and proportions and body fat distribution.
2. To determine changes in genome-wide gene expression and DNA methylation profiles related to insulin sensitivity in fat, muscle and endometrial tissue biopsies, and biomarkers in whole blood.
3. To evaluate endocrine measures including menstrual pattern and ovulation frequency, circulating hormones (sex steroids, AMH, gonadotropins), and excretion of metabolites of sex steroids in urine.
4. To determine changes in women's HRQoL, symptoms of anxiety and depression, dieting and eating patterns, and negative side-effects.
5. To evaluate the cost-effectiveness of the different treatments.

ELIGIBILITY:
Inclusion criteria - women with PCOS:

1. Age 18 to 40 years
2. Body mass index (BMI) ≥25 to ≤40 given that 95% of all women with PCOS with a BMI ≥25 are insulin resistant (71,72).
3. PCOS diagnosis according to Rotterdam criteria 2003 (73), with at least two of the following three symptoms: Clinical signs of hyperandrogenism (hirsutism or acne); oligo/amenorrhea; and/or polycystic ovaries (PCOS). Hirsutism is defined as a self-reported Ferriman-Gallwey (FG) score ≥8 (≥5 Asian) (74,75). Acne is defined by a positive response to the question Do you have acne? Oligomenorrhea is defined as an intermenstrual interval >35 days and <8 menstrual bleedings in the past year. Amenorrhea as <3 cycles per year. PCO is defined by transvaginal ultrasound with ≥12 follicles 2-9 mm and/or ovarian volume ≥10 ml in one or both ovaries.
4. Willing to sign the consent form.

Inclusion criteria - controls:

Controls should have BMI >25 to <40, regular cycles with 28 days ± 2 days, and no signs of hyperandrogenism. They are excluded if they have menstrual irregularities, signs of hyperandrogenism (FG >4), or evidence of PCO morphology on ultrasound.

Exclusion criteria for all women

1. Age >40
2. Exclusion of other endocrine disorders such as non-classic congenital adrenal hyperplasia (17-hydroxyprogesterone < 3nmol/L), androgen secreting tumors or suspected Cushing's syndrome.
3. Having known renal disease (creatinine clearance < 60 mL/min), hepatic insufficiency, autoimmune disorders or cancer.
4. Any acute condition with potential to alter renal function or cause tissue hypoxia.
5. Type I diabetes.
6. Pharmacological treatment (cortizon, antidepressant, other antidiabetic treatment such as insulin and acarbose, hormonal contraceptives, hormonal ovulation induction or other drugs judged by discretion of investigator) within 12 weeks. Depo Provera or similar within 6 months.
7. Hypersensitivity to metformin hydrochloride or to any of the excipients.
8. Blood pressure >160 / 100 mmHg
9. Pregnancy or breastfeeding the last 6 months
10. Acupuncture the last 2 months
11. Daily smoking and alcoholic intake
12. Language barrier or disabled person with reduced ability to understand the information given.

In total 50 controls will be matched at baseline (age, weight and BMI) to women with PCOS. Controls will undergo screening and baseline visit, but will not be randomized to any treatment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 303 (Estimated)
Dates: Start 2015-12; Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to after 4 months in HOMA-IR [fasting insulin (μU/mL) × fasting glucose (mmol/L)] / 22.5) | 4 months
  Changes from baseline to after 4 months of treatment in HOMA-IR [fasting insulin (μU/mL) × fasting glucose (mmol/L)] / 22.5) between 1) acupuncture + lifestyle management and 2) metformin + lifestyle management compared to 3) lifestyle management only.
Changes from baseline to after 4 months of treatment in HbA1c | 4 months
  Changes from baseline to after 4 months of treatment in HbA1c between 1) acupuncture + lifestyle management and 2) metformin + lifestyle management compared to 3) lifestyle management only.
Changes from baseline to after 4 months of treatment in insulin response to glucose during the oral glucose tolerance test (OGTT) | 4 months
  Changes from baseline to after 4 months of treatment in insulin response to glucose during the OGTT (AUC using the trapezoidal rule) between 1) acupuncture + lifestyle management and 2) metformin + lifestyle management compared to 3) lifestyle management only.

SECONDARY OUTCOMES:
Changes from baseline to after 4 months and again 4 months after last treatment in secondary metabolic measures | 8 months
  Changes in secondary metabolic measures with calculation of e.g. HOMA-B
Changes from baseline to after 4 months and again 4 months after last treatment gene expression and DNA methylation profiles related to insulin sensitivity in fat, muscle and endometrial tissue biopsies, and biomarkers in whole blood. | 8 months
  Changes in mRNA gene expression and DNA methylation expression and biomarkers in whole blood.
Changes from baseline to after 4 months and again 4 months after last treatment in menstrual pattern. | 8 months
  Changes in menstrual pattern per month.
Changes from baseline to after 4 months and again 4 months after last treatment in circulating reproductive hormones. | 8 months
  Changes in circulating circulating reproductive hormones.
Changes from baseline to after 4 months and again 4 months after last treatment in women's HRQoL. | 8 months
  Changes in women's HRQoL measured with polycystic ovary syndrome questionnaire (PCOSQ) and short form-36 (SF36) two validated questionnairs.
Changes from baseline to after 4 months and again 4 months after last treatment in women's symptoms of anxiety and depression. | 8 months
  Changes in women's symptoms of anxiety and depression measured with the self-reported version of the Comprehensive Psychopathological Rating Scale for Affective Syndromes (CPRS-S-A).
Changes from baseline to after 4 months and again 4 months after last treatment in women's dieting and eating patterns. | 8 months
  Changes in women's dieting and eating patterns assessed with Three-Factor Eating Questionnaire (TFEQ-R21), and Questionnaire of Eating and Weight Patterns-Revised (QEWP-R).
Cost-effectiveness of the different treatments throughout the study. | 8 months
  Cost-effectiveness of the different treatments by calculation of e.g. treatment visits, time for patient and with EuroQol-5 dimension (EQ-5D).

CONTACTS AND LOCATIONS:
Overall Officials: Elisabet Stener-Victorin, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Peking University, Beijing, China
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stener-Victorin E, Zhang H, Li R, Friden C, Li D, Wang W, Wang H, Chang C, Li S, Huo Z, Zhang H, Ji X, Linden-Hirschberg A, Qiao J. Acupuncture or metformin to improve insulin resistance in women with polycystic ovary syndrome: study protocol of a combined multinational cross sectional case-control study and a randomised controlled trial. BMJ Open. 2019 Jan 4;9(1):e024733. doi: 10.1136/bmjopen-2018-024733. PMID 30612112